CLINICAL TRIAL: NCT06542549
Title: Efficacy and Safety of AK104 (PD-1/CTLA-4 Bi-specific Antibody) Combined With Chemotherapy for Neoadjuvant Treatment of Advanced Ovarian Cancer: a Randomized Controlled, Single-center Clinical Study
Brief Title: Efficacy and Safety of AK104 (PD-1/CTLA-4 Bispecial Antibody) Combined With Chemotherapy for Neoadjuvant Treatment of Advanced Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhouYing-Remat
Record Dates: First submitted 2024-07-28; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Advanced Ovarian Cancer; AK104(PD-1/CTLA-4 Bispecial Antibody); Chemotherapy; Efficacy; Safety

STUDY DESIGN:
Intervention Model Description: Subjects in the experimental group received AK104 combined chemotherapy for 3-4 cycles (determined by the investigator) before surgery, and subjects in the control group received chemotherapy for 3-4 cycles (determined by the investigator) before surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK104 combined with chemotherapy (Experimental): 10mg/kg, administered every three weeks. The drug was administered by intravenous infusion for 60 minutes (±10 minutes). For subjects who cannot tolerate a 60-minute infusion, the infusion time can be extended up to 120 minutes. Dose adjustment is not allowed during treatment; Delayed dosing is allowed.
  Interventions: Drug: AK104
- chemotherapy only (No Intervention): Conventional chemotherapy regimen can be selected: ① Paclitaxel: 175mg/㎡, intravenous infusion d1+ carboplatin AUC5, intravenous infusion d1, Q3W; ② Paclitaxel (albumin-bound type) 260mg/m2 d1+ carboplatin AUC 5, d1, Q3W; (Limited to patients who are allergic to solvent-based paclitaxel solute (polyoxyethylene castor oil) or to paclitaxel/docetaxel, paclitaxel (albumin-bound type) can be substituted in the combination regimen), ③ paclitaxel (albumin-bound type) 260mg/m2 d1+ cisplatin: 75mg/m2 d1, Q3W. (Limited to patients who are allergic to solvent-based paclitaxel solutes (polyoxyethylene castor oil) or to paclitaxel/docetaxel, paclitaxel (albumin-bound) can be substituted in the combination regimen)

INTERVENTIONS:
Drug: AK104 — The study treatment was followed by a 3-week treatment cycle. The dosing time window is ±3 days. Within 72 hours before each dosing cycle, subjects are required to complete various examinations, including vital signs, physical examination, laboratory examination, and physical status score, to evaluate the safety and tolerability of continued treatment.
  Arms: AK104 combined with chemotherapy

SUMMARY:
This is a randomized, controlled, single-center clinical study to evaluate AK104 in FIGO 2018 stage III-IV ovarian cancer subjects who were assessed to be at high perioperative risk and/or unable to achieve R0 resection prior to initial treatment. The efficacy and safety of neoadjuvant therapy with intravenous infusion combined with chemotherapy compared with chemotherapy alone.

DETAILED DESCRIPTION:
Subjects in the experimental group received AK104 combined chemotherapy for 3-4 cycles (determined by the investigator) before surgery, and subjects in the control group received chemotherapy for 3-4 cycles (determined by the investigator) before surgery. Treatment until unless intolerable toxicity occurs, informed consent is withdrawn, or other criteria for discontinuation are met.

The study treatment was followed by a 3-week treatment cycle. The dosing time window is ±3 days. Within 72 hours before each dosing cycle, subjects are required to complete various examinations, including vital signs, physical examination, laboratory examination, and physical status score, to evaluate the safety and tolerability of continued treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to sign the informed consent form.
2. 18 years ≤ age <75 years, female.
3. Patients with epithelial ovarian cancer (high-grade serous adenocarcinoma, ovarian endometrial carcinoid adenocarcinoma), peritoneal or fallopian tube carcinoma, or clear cell carcinoma confirmed by histopathology, FIGO 2018 stage III-IV.
4. Evidence of compliance with neoadjuvant chemotherapy for ovarian cancer: (a) Preoperative evaluation by gynecologic oncologists (multidisciplinary if necessary) indicates that R0 resection is less likely to be achieved after primary tumor reduction; (b) Patients whose physical state cannot tolerate PDS and are not suitable for immediate surgery (such as perioperative high risk, old age, medical complications, etc.); (c) Without any systematic anti-tumor therapy for ovarian cancer (including but not limited to radiotherapy, chemotherapy, surgery, targeted therapy and immunotherapy); Note: Histopathology is obtained by puncture biopsy, laparoscopic exploration, etc. Lymph node resection or biopsy for clinical staging purposes is permitted.
5. Those with at least one measurable lesion (RECIST version 1.1).
6. ECOG Physical status score 0-2.
7. Estimated survival time > 12 weeks.
8. Good organ function.
9. Participants of reproductive age must agree to use effective contraception during the trial; Serum or urine pregnancy tests for women of childbearing age must be negative.
10. Non-lactating patients.

Exclusion Criteria:

1. Ovarian cancer, fallopian tube cancer, primary peritoneal cancer (such as germ cell tumor) of non-epithelial origin; Ovarian tumors with low malignant potential (e.g., borderline tumors).
2. Patients with other malignant tumors in the past (within 5 years) or at the same time, with the exception of cured local tumors (such as basal cell skin cancer, squamous cell skin cancer, superficial bladder cancer, cervical carcinoma in situ, breast carcinoma in situ, etc.) and breast cancer with no recurrence >3 years after radical surgery.
3. Subjects with active viral hepatitis B, inactive or asymptomatic hepatitis B virus (HBV) carriers (HBV surface antigen [HBsAg] positive) with HBV DNA > 1000 IU/mL, and subjects with active viral hepatitis C. Note: Inactive or asymptomatic carriers, treated and stable hepatitis B subjects with HBV DNA ≤ 1000 IU/mL were admitted. Subjects with cured viral hepatitis C, HCVAb positive and HCV RNA negative were admitted.
4. A history of testing positive for known human immunodeficiency virus or known acquired immunodeficiency syndrome.
5. Have an active or possibly recurring autoimmune disease; The following are excluded: vitiligo, alopecia, psoriasis or eczema that do not require systematic treatment; Hypothyroidism due to autoimmune thyroiditis requires only stable dose hormone replacement therapy; Only a steady dose of insulin replacement is required for type 1 diabetes.
6. A history of severe allergic reactions to any monoclonal antibody and/or investigational drug ingredient.
7. Subjects with known active TB and suspected active TB should undergo clinical examination to rule out known active syphilis infection.
8. There is a history or current presence of noninfectious pneumonia/interstitial lung disease requiring systemic glucocorticoid therapy.
9. Severe infections occurring within 4 weeks prior to first dosing, including but not limited to active infections with comorbidification requiring hospitalization, sepsis, or severe pneumonia that received systemic anti-infective therapy within 2 weeks prior to first dosing (excluding antiviral therapy for hepatitis B or C).
10. Serious medical conditions or concomitant non-oncological conditions, such as neurological disorders, psychosis, infectious diseases, or laboratory abnormalities, may increase the risk of participating in the study or taking the investigational drug, which the investigator believes would make the patient unfit for entry into the study.
11. Patients with clinically significant cardiovascular disease.
12. Patients who were judged by the investigator to be unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
R0 rate | Up to 6 months
  Rate of complete tumor resection (R0): complete resection of the visible lesion.

SECONDARY OUTCOMES:
ORR | 1 year
  Objective tumor response rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as best overall response according to radiological assessments.
DCR | 1 year
  Disease control rate (DCR) refers to the percentage of cases with remission and disease stability after treatment in the total number of evaluable cases.
pCR | 1 year
  Pathological complete response is the breast primary focus and axillary lymph node surgery specimen pathological examination without invasive tumor cell residual.
PFS | 1 year
  Progress free survival is defined as the length of time from random assignment to disease progression or to death resulting from any cause other than the progress.
AE | 1 year
  adverse events are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.